CLINICAL TRIAL: NCT00635999
Title: Desensitization and Cognitive Therapy in General Anxiety
Brief Title: A Comparison Between Cognitive, Behavioral, and Cognitive-Behavioral Therapy for Generalized Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michelle G. Newman (Other)
Responsible Party: Sponsor-Investigator, Michelle G. Newman, Study Director, Penn State University
Organization: Penn State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH039172-01 (NIH)
Record Dates: First submitted 2008-03-12; First posted 2008-03-14 (Estimated); Results first posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Purely Behavioral therapy (Experimental): Participants will receive treatment with progressive and applied relaxation and self-control desensitization.
  Interventions: Behavioral: Applied relaxation and self-control desensitization
- Cognitive-Behavioral Therapy (Experimental): Participants will receive treatment with cognitive therapy, progressive and applied relaxation, and self-control desensitization
  Interventions: Behavioral: Cognitive-Behavioral Therapy
- Cognitive Therapy (CT) (Experimental): Participants will receive purely cognitive therapy including identification of maladaptive thought processes and training in cognitive restructuring.
  Interventions: Other: Cognitive therapy (CT)

INTERVENTIONS:
Behavioral: Applied relaxation and self-control desensitization — Applied relaxation and self-control desensitization sessions will teach participants relaxation techniques and the use of imagery for coping with anxiety. Treatment will include 14 weekly sessions.
  Arms: Purely Behavioral therapy
Other: Cognitive therapy (CT) — CT sessions will teach participants to identify ways in which they perceive themselves and the world and how to modify these thoughts to reduce anxiety. CT will include 14 weekly sessions.
  Arms: Cognitive Therapy (CT)
Behavioral: Cognitive-Behavioral Therapy — Includes all of the techniques in the other 2 interventions.
  Arms: Cognitive-Behavioral Therapy

SUMMARY:
This study will evaluate the effectiveness of three adaptive coping treatments in lessening anxiety in adults with generalized anxiety disorder.

DETAILED DESCRIPTION:
Generalized anxiety disorder (GAD) is a common psychiatric disorder that affects nearly 6.8 million adults in the United States. GAD is characterized by persistent feelings of worry and anxiety that remain even when there is little reason for concern. The excessive worry that people with GAD experience can be so extreme that carrying out activities of daily life becomes difficult. GAD is often accompanied by physical symptoms as well, including muscle aches, nausea, sweating, exhaustion, irritability, frequent urination, and shaking. People with GAD are also at a higher risk for other disorders, including depression and substance abuse, making early treatment of GAD important. Forms of psychotherapy that concentrate on stress management, relaxation techniques, and control of thoughts about anxiety-provoking situations may be effective treatments for people with GAD. This study will evaluate the effectiveness of three adaptive coping treatments, relaxation and self-control desensitization, cognitive behavioral therapy (CBT), and a combination of the two, in lessening anxiety in adults with GAD.

Participation in this study will last about 28 months. All participants will first complete three assessment sessions that will include an interview about anxiety symptoms and medical history, self-report questionnaires, and a physiological evaluation. After the first interview, participants will be asked to rate their level of anxiety four times a day in a diary. They will continue with these daily diary entries through the completion of treatment. Once participants complete the first 2 weeks' worth of daily ratings, participants will be assigned randomly to receive treatment with relaxation and self-control desensitization, CBT, or a combination of the two treatments. All participants will receive 14 weekly treatment sessions lasting between 1.5 and 2 hours each. During CBT sessions, participants will learn to identify ways in which they perceive themselves and the world and how to modify these thoughts to reduce anxiety. Applied relaxation and self-control desensitization sessions will teach participants relaxation techniques and the use of imagery for coping with anxiety. Between sessions, all participants will complete homework assignments that will involve practicing the approaches learned in sessions and continuing the daily diaries.

Upon completion of treatment, participants will repeat the initial assessments. Follow-up visits will occur at Months 6, 12, and 24 after treatment completion and will include repeat interview and self-report sessions and completion of 1 week's worth of daily diary entries before each visit.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of GAD

Exclusion Criteria:

* Diagnosis of any of the following: panic disorder, subclinical GAD, severe depression, psychosis, or organic brain syndrome
* Currently receiving therapy for GAD or has previously received CBT
* Medical contributions to anxiety
* Currently taking antidepressant medication
* Current substance abuse

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 1991-10; Primary Completion 1998-10 (Actual); Study Completion 1998-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle G. Newman, PhD, Study Director — Penn State University; Thomas D. Borkovec, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Summary data has been shared.

REFERENCES:
- [Background] Roemer L, Molina S, Borkovec TD. An investigation of worry content among generally anxious individuals. J Nerv Ment Dis. 1997 May;185(5):314-9. doi: 10.1097/00005053-199705000-00005. PMID 9171808
- [Background] Roemer L, Molina S, Litz BT, Borkovec TD. Preliminary investigation of the role of previous exposure to potentially traumatizing events in generalized anxiety disorder. Depress Anxiety. 1996-1997;4(3):134-8. doi: 10.1002/(SICI)1520-6394(1996)4:33.0.CO;2-G. PMID 9166642
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Schut AJ, Castonguay LG, Borkovec TD. Compulsive checking behaviors in generalized anxiety disorder. J Clin Psychol. 2001 Jun;57(6):705-15. doi: 10.1002/jclp.1043. PMID 11344459
- [Background] Stöber, J., & Borkovec, T. D. (2002). Reduced concreteness of worry in generalized anxiety disorder: Findings from a therapy study. Cognitive Therapy and Research, 26, 89-96.
- [Background] Behar E, Alcaine O, Zuellig AR, Borkovec TD. Screening for generalized anxiety disorder using the Penn State Worry Questionnaire: a receiver operating characteristic analysis. J Behav Ther Exp Psychiatry. 2003 Mar;34(1):25-43. doi: 10.1016/s0005-7916(03)00004-1. PMID 12763391
- [Background] McLaughlin KA, Behar E, Borkovec TD. Family history of psychological problems in generalized anxiety disorder. J Clin Psychol. 2008 Jul;64(7):905-18. doi: 10.1002/jclp.20497. PMID 18509873
- [Background] Cassidy J, Lichtenstein-Phelps J, Sibrava NJ, Thomas CL Jr, Borkovec TD. Generalized anxiety disorder: connections with self-reported attachment. Behav Ther. 2009 Mar;40(1):23-38. doi: 10.1016/j.beth.2007.12.004. Epub 2008 Jun 24. PMID 19187814
- [Background] Newman MG, Przeworski A, Fisher AJ, Borkovec TD. Diagnostic comorbidity in adults with generalized anxiety disorder: impact of comorbidity on psychotherapy outcome and impact of psychotherapy on comorbid diagnoses. Behav Ther. 2010 Mar;41(1):59-72. doi: 10.1016/j.beth.2008.12.005. Epub 2009 Jun 8. PMID 20171328
- [Background] Newman MG, Fisher AJ. Expectancy/Credibility Change as a Mediator of Cognitive Behavioral Therapy for Generalized Anxiety Disorder: Mechanism of Action or Proxy for Symptom Change? Int J Cogn Ther. 2010 Sep;3:245-261. doi: 10.1521/ijct.2010.3.3.245. PMID 21132075
- [Result] Borkovec TD, Newman MG, Pincus AL, Lytle R. A component analysis of cognitive-behavioral therapy for generalized anxiety disorder and the role of interpersonal problems. J Consult Clin Psychol. 2002 Apr;70(2):288-98. PMID 11952187

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Principal diagnosis of GAD, no panic disorder, Clinician's Severity Rating (CSR) for GAD of 4 or more, absence of concurrent therapy, no history of having received CBT methods in prior therapy, no medical contributions to the anxiety, no antidepressant medication, and absence of severe MDD, substance abuse, psychosis, and organic brain syndrome.
Groups:
- Self-control Desensitization: Participants will receive treatment with applied relaxation and self-control desensitization.
- Cognitive Therapy: Participants will receive treatment with cognitive therapy.
- Combined Cognitive Behavioral Therapy: Participants will receive treatment with a combination of applied relaxation, self-control desensitization, and cognitive behavioral therapy.
Period: Overall Study
Arm/Group | Self-control Desensitization | Cognitive Therapy | Combined Cognitive Behavioral Therapy
Started | 27 | 25 | 24
Completed | 23 | 23 | 23
Not Completed | 4 | 2 | 1
Not completed — Withdrawal by Subject | 4 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-control Desensitization | Cognitive Therapy | Combined Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 27 | 25 | 24 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 25 | 24 | 76
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.02 (10.36) | 38.42 (11.10) | 35.64 (13.92) | 37.36 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 16 | 52
  Male | 8 | 8 | 8 | 24
Region of Enrollment [Number; unit: participants]
  United States | 27 | 25 | 24 | 76

OUTCOME MEASURES:

1. Primary Outcome: High End State Function
Description: Percentage of participants meeting high end state functioning (e.g., within 1 standard deviation of mean of nonanxious samples on Hamilton Anxiety Rating Scales, Spielberger's State-Trait Anxiety Inventory, Penn State Worry Questionnaire, and Reactions to Relaxation and Arousal Questionnaire)
Time Frame: 10-14 days after last therapy session and months 6, 12, and 24 following last therapy session
Population: People who completed treatment
Measure: Number; unit: % people meeting high endstate status
Arm/Group | Self-control Desensitization | Cognitive Therapy | Combined Cognitive Behavioral Therapy
Number analyzed (Participants) | 23 | 23 | 23
% people meeting high endstate status
  10-14 days after last therapy session | 56.52 | 43.48 | 56.52
  6 month follow-up | 47.62 | 68.18 | 56.52
  12 month follow-up | 28.57 | 47.62 | 43.48
  24 month follow-up | 47.62 | 52.38 | 38.10

2. Secondary Outcome: Within-group Change Represented as Cohen's d Effect Sizes
Description: Cohen's d within-group effect sizes comparing pre-therapy assessment to assessment at 10-14 days after last therapy session, at 6-month follow-up, at 12-month follow-up, and at 24-month follow-up. Findings reported in table are Cohen's d effect sizes averaged over Hamilton Anxiety Scale (scores ranging from 0-56, higher scores mean more anxiety), the Assessor Severity Scale (scores ranging from 0-8, higher scores mean more severity), and the State-Trait Anxiety Inventory-Trait version (scores ranging from 20-80, higher scores mean more state anxiety). The within-group effective sizes are the posttherapy [or follow-up] mean minus pretherapy mean divided by the pretherapy standard deviation.
Time Frame: 10-14 days after last therapy session and months 6, 12, and 24 following last therapy session
Population: People who completed treatment
Measure: Number; unit: Cohen's d within group effect size
Arm/Group | Self-control Desensitization | Cognitive Therapy | Combined Cognitive Behavioral Therapy
Number analyzed (Participants) | 23 | 23 | 23
Cohen's d within group effect size
  10-14 days after last therapy session | 2.38 | 2.95 | 2.8
  6 month follow-up | 2.35 | 2.81 | 2.86
  12 month year follow-up | 2.43 | 2.48 | 2.45
  24 month follow-up | 2.34 | 2.67 | 2.31

ADVERSE EVENTS:
Arm/Group | Self-control Desensitization | Cognitive Therapy | Combined Cognitive Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes